CLINICAL TRIAL: NCT03867253
Title: A Multicentre,Randomised, Double-blind, Placebo-controlled, 3-arm, 24-week Parallel-group Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of ORY-2001 in Patients With Mild-moderate Alzheimer's Disease
Brief Title: Testing the Safety and Preliminary Efficacy of the New Drug ORY-2001 in Mild to Moderate Alzheimer's Disease
Acronym: ETHERAL-US
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oryzon Genomics S.A. (Industry)
Collaborators: Alzheimer's Drug Discovery Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL05-ORY-2001US
Record Dates: First submitted 2019-02-20; First posted 2019-03-07 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2020-07

CONDITIONS: Mild to Moderate Alzheimer's Disease
Keywords: Alzheimer's Disease, ORY-2001
MeSH Terms: conditions — Alzheimer Disease | interventions — vafidemstat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ORY-2001 Low dose (Active Comparator): 0.6mg ORY-2001 capsule
  Interventions: Drug: ORY-2001 Low dose
- ORY-2001 High dose (Active Comparator): 1.2mg ORY-2001 capsule
  Interventions: Drug: ORY-2001 High dose
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ORY-2001 Low dose — 0.6mg ORY-2001 capsule
  Arms: ORY-2001 Low dose
Drug: ORY-2001 High dose — 1.2mg ORY-2001 capsule
  Arms: ORY-2001 High dose
Drug: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
This is a Phase IIa study assessing the safety, tolerability and preliminary efficacy of ORY-2001 in mild to moderate Alzheimer's Disease patients.

DETAILED DESCRIPTION:
This phase IIa study is a double-blind, randomized, parallel-group and multicenter study with a placebo-controlled 24-week treatment period followed by a no placebo-controlled 24-week extension period.

It is planned to randomise 25 patients. In the double-blind placebo-controlled treatment period, all patients will be randomized between two doses of ORY-2001 and placebo. In the double-blind no placebo-controlled extension period, patients in the placebo arm will be re-allocated in one of the two different dose levels of ORY-2001. Randomization will be stratified by cognitive impairment severity.

An independent Data Monitoring Committee (DMC) will review un-blinded safety data throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Probable Alzheimer's Disease (AD) diagnosed according to National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
* MMSE score at Screening and Baseline Visits of at least 16 and not greater than 26
* Evidence of the AD pathophysiological process indicated by decreased levels of amyloid antigen binding (AB) and increased levels of total Tau protein or phospho-Tau protein in cerebrospinal fluid (CSF)
* Outpatient consulting a general practitioner, or a psychiatrist/neurologist/geriatrician
* Knowledgeable and reliable close relative/caregiver who will accompany the patient to all clinic visits during the study
* Daily treatment with the same acetylcholinesterase inhibitor on a stable dose
* Fertile male and female must use highly effective contraception, from the Screening Visit until 90 days after last dose.
* Signed informed consent by patient (or legal representative, if applicable) and a close relative/caregiver prior to the initiation of any study specific procedure

Exclusion Criteria:

* Failure to perform screening or baseline examinations
* Hospitalization or change of concomitant medication 1 month prior to Screening visit or during Screening Period
* Clinical, laboratory or neuroimaging findings consistent with:

  1. Other primary degenerative dementia;
  2. Other neurodegenerative condition;
  3. Cerebrovascular disease;
  4. Other central nervous system diseases;
* A current Diagnostic and Statistical Manual-5 (DSM-5) diagnosis of major depression, schizophrenia or bipolar disorder
* Positive results for tuberculosis, human immunodeficiency virus (HIV), hepatitis C or hepatitis B (hepatitis B surface antigen [HbsAg]) serology at the Screening Visit
* Clinically significant, advanced or unstable disease that may interfere with evaluation.
* Disability that may prevent the patients from completing all study requirements.
* Chronic drug intake of forbidden concomitant medication.
* Treatment with anti-amyloid beta or anti-Tau protein monoclonal antibodies or other disease modifying strategies within three months or five half-lives, whichever is longer, prior to the Screening Visit
* Treatment with an active vaccine targeting amyloid beta or Tau protein
* Suspected or known drug or alcohol abuse
* Metallic implants or any other cause precluding the performance of brain MRI
* Enrolment in another investigational study or intake of investigational drug within the previous 3 months since the last dose
* Suicide attempt within the last year or significant risk of suicide (in the opinion of the investigator, defined as a "yes" to suicidal ideation questions 4 or 5, or answering "yes" to suicidal behavior on the Columbia-Suicide Severity Rating Scale within the past 12 months)
* Any condition that in the opinion of the investigator makes the patient unsuitable for inclusion in the study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events | Week 24
  Number, frequency and severity of Treatment Emergent Adverse Events (TEAEs) including serious TEAEs.
Treatment Emergent Adverse Events | Week 48
  Number, frequency and severity of Treatment Emergent Adverse Events (TEAEs) including serious TEAEs.
Withdrawn patients due to TEAEs | Week 24
  Number and percentage of withdrawn patients due to TEAEs
Withdrawn patients due to TEAEs | Week 48
  Number and percentage of withdrawn patients due to TEAEs

SECONDARY OUTCOMES:
Cohen-Mansfield Agitation Inventory (CMAI) | 48 weeks
  Change from baseline to week 48 compared to placebo
Clinician version of the Apathy Evaluation Scale (AES-C) | 48 weeks
  Change from baseline to week 48 compared to placebo
14-item Alzheimer's Disease Assessment Scale-Cognitive | 48 weeks
  Change from baseline to week 48 compared to placebo
Computerized Cognitive Test battery | 48 weeks
  Change from baseline to week 48 compared to placebo
Mini-Mental State Examination (MMSE) | 48 weeks
  Change from baseline compared to placebo
Clinical Dementia Rating Scale Sum of Boxes | 48 weeks
  Change from baseline to week 48 compared to placebo
Cornell Scale for Depression in Dementia (CSDD) | 48 weeks
  Change from baseline to week 48 compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ropacki, MD, Study Director — Oryzon Genomics S.A.
Locations (4):
- United States (4):
  - Alzheimer's Research and Treatment Center, Wellington, Florida
  - Columbus Memory Center, Columbus, Georgia
  - Princeton Medical Institute, Princeton, New Jersey
  - Abington Neurological Associates Ltd., Willow Grove, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided